CLINICAL TRIAL: NCT01063751
Title: A Prospective, Post-market, Multi-center Study of the Tritanium® Acetabular Shell
Brief Title: Tritanium® Primary Acetabular Shell Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: As longitudinal patient follow-up continues to lag, Stryker has determined that the study is no longer able to meet the regulatory requirements this study intends to support.
  Termination is not related to any safety concerns with the products.
Sponsor: Stryker Orthopaedics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 69
Record Dates: First submitted 2010-02-04; First posted 2010-02-05 (Estimated); Results first posted 2024-01-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2024-12

CONDITIONS: Arthroplasty, Replacement, Hip
Keywords: Osteoarthritis; Traumatic arthritis; Avascular Necrosis
MeSH Terms: conditions — Osteoarthritis; Osteonecrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tritanium® Primary Acetabular Shell (Other): Tritanium® Primary Acetabular Shell
  Interventions: Device: Tritanium® Primary Acetabular Shell

INTERVENTIONS:
Device: Tritanium® Primary Acetabular Shell — Tritanium® Primary Acetabular Shell in total hip replacement.

SUMMARY:
This study will be a prospective, non-randomized evaluation of the Tritanium® Acetabular Shell for primary total hip replacement (THR) with a cementless application in a consecutive series of patients who meet the eligibility criteria. Half of the cases will use the Trident® X3® polyethylene insert alone as the bearing surface; the other half will use the modular dual mobility (MDM™) liner coupled with a compatible anatomic dual mobility (ADM™)/MDM™ X3® insert as the bearing surface.

The success rate, defined as freedom from acetabular revision for any reason, for hips implanted with the Tritanium® Acetabular Shell, is no worse than for hips implanted with similar technology as reported in the literature and Trident® X3® Study historical control at 5 years postoperative.

DETAILED DESCRIPTION:
The Tritanium® Acetabular Shell, cleared for use under FDA 510(k) K081171, is a hemispherical acetabular shell with a 3D surface for biological fixation, fabricated from Commercially Pure Titanium (CPTi). The shell is built upon the design features and clinical history of the existing Trident® Tritanium®, Trident® AD, and Trident® hemispherical acetabular (HA) shells. The device is designed with a roughened surface and high coefficient of friction to resist micromotion and promote initial fixation. The Tritanium® Acetabular Shell, intended for use in a cementless application, is available in sizes from 44 millimeter (mm) through 66 mm and is compatible with Trident® polyethylene insert and acetabular screws. This advanced technology is designed to address the need for improved initial and biological fixation. Data in support of these marketing claims will be collected in the Tritanium® Primary Acetabular Shell Study.

A prospective, post-market, multi-center design will be employed. Radiographs will be assessed by an independent reviewer.

Cases will be enrolled at 7 to 12 centers. The enrollment goal ranges from 20 to 34 cases implanted with the Tritanium® Acetabular Shell per center. The enrollment goal range is dependent upon the number of participating centers as well as the relative rates of enrollment of the two treatment groups. Although a range is presented, there is no maximum limit to the number of cases that a center may enroll. In the event that a center far exceeds the overall enrollment goal or enrollment into one of the treatment groups is completed, Stryker may ask the center to cease enrollment so as not to skew the data. All participating centers will comply with the federal regulations regarding patient informed consent and Institutional Review Board (IRB) approval. Non-compliance of a study center may result in termination of the center's participation in the study.

ELIGIBILITY:
Inclusion Criteria:

* A. Patient has signed an IRB approved, study specific Informed Patient Consent Form.
* B. Patient is a male or non-pregnant female age 18 years or older at time of study device implantation.
* C. Patient has primary diagnosis of Non-Inflammatory Degenerative Joint Disease (NIDJD).
* D. Patient is a candidate for a primary cementless total hip replacement.
* E. Patient is willing and able to comply with postoperative scheduled clinical and radiographic evaluations and rehabilitation.

Exclusion Criteria:

* F. Patient has a Body Mass Index (BMI) ≥ 40.
* G. Patient has an active or suspected latent infection in or about the affected hip joint at time of study device implantation.
* H. Patient has a neuromuscular or neurosensory deficiency, which limits the ability to evaluate the safety and efficacy of the device.
* I. Patient is diagnosed with a systemic disease (e.g. Lupus Erythematosus) or a metabolic disorder (e.g. Paget's Disease) leading to progressive bone deterioration.
* J. Patient is immunologically suppressed or receiving steroids in excess of normal physiological requirements (e.g. > 30 days).
* K. Patient requires revision surgery of a previously implanted total hip replacement or hip fusion to the affected joint.
* L. Patient has a known sensitivity to device materials.
* M. Patient is a prisoner.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 275 (Actual)
Dates: Start 2011-07; Primary Completion 2022-05-05 (Actual); Study Completion 2023-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Kopko, MD, Principal Investigator — Syracuse Orthopedic Specialists, P.C.; John Noble, MD, Principal Investigator — Center for Orthopaedics and Spine, LLP; Carmen Crofoot, MD, Principal Investigator — Northern Light Eastern Maine Medical Center; John Diana, MD, Principal Investigator — Adventist Health St. Helena; Stephen Duncan, MD, Principal Investigator — University of Kentucky Research Foundation; Brock Lindsey, MD, Principal Investigator — West Virginia University; Stephen Raterman, MD, Principal Investigator — Florida Medical Clinic
Locations (7):
- United States (7):
  - Adventist Health St. Helena, St. Helena, California
  - Florida Medical Clinic, Tampa, Florida
  - University of Kentucky Research Foundation, Lexington, Kentucky
  - Center for Orthopaedics and Spine, LLP, Lake Charles, Louisiana
  - Northern Light Eastern Maine Medical Center, Bangor, Maine
  - Syracuse Orthopedic Specialists, P.C., Syracuse, New York
  - West Virginia University, Morgantown, West Virginia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 275 participants/284 hip cases were enrolled. There were 266 unilateral hip cases and 9 bilateral hips cases.
Units Other Than Participants: Hips
Period: Overall Study
Arm/Group | Tritanium® Primary Acetabular Shell
Started | 275; 284 Hips (275 subjects were enrolled making up 284 hip cases. There were 266 unilateral hip cases and 9 bilateral hips cases)
Completed | 41; 43 Hips (1 bilateral participant had 1 case/hip which completed the study and 1 case/hip which was censored from the study analyses. This participant is being included in the "Completed" category and will not be included in the "Censored from analyses" category.)
Not Completed | 234; 241 Hips
Not completed — Censored from analyses | 42
Not completed — Withdrawal by Subject | 34
Not completed — Lost to Follow-up | 30
Not completed — Death | 13
Not completed — Sponsored Terminated Study | 60
Not completed — Cases terminated due to investigator leaving the site and site closure. | 35
Not completed — Investigator site closed | 10
Not completed — Revision | 6
Not completed — Physician Decision | 4

BASELINE CHARACTERISTICS:
Population: 275 participants were enrolled making up 284 hip cases. Of the 284 hips, 43 cases were censored and not included in the data analyses. Therefore, 241 cases were included in the analyses.
  Of the 284 cases/234 participants, 42 cases completed the study per protocol. 40 participants made up these 42 cases.
Units Other Than Participants: hips
Arm/Group | Tritanium® Primary Acetabular Shell
Number analyzed (Participants) | 234
Number analyzed (hips) | 241
Age, Continuous [Mean (Full Range); unit: years] — For bilateral total knee replacement participants, the age at the time of initial knee replacement surgery is used.
  years | 62.60 [31 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100
  Male | 134
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 21
  White | 207
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: Cases]
  United States | 241

OUTCOME MEASURES:

1. Primary Outcome: Absence of Acetabular Revision
Description: To evaluate the success rate of cementless primary total hip replacement (THR) in hips implanted with the Tritanium® Acetabular Shell, as compared to the published results of similar acetabular components. Success will be defined as absence of acetabular shell revision for any reason at 5 years postoperative. It is expected that the survivorship of the Tritanium® Acetabular Shell group will be non-inferior to the survivorship reported in the literature for similar competitive devices.
Time Frame: 5 years
Measure: Count of Units; unit: hips
Units Other Than Participants: hips
Arm/Group | Tritanium® Primary Acetabular Shell
Number analyzed (Participants) | 234
Number analyzed (hips) | 241
hips | 6

2. Secondary Outcome: Rates of Screw Fixation Usage in the Tritanium® Acetabular Shell
Description: Usage of bone screw fixation will be recorded and compared between the Tritanium® Acetabular Shell group and the Trident® Hemispherical Acetabular (HA) Shell group (Trident® X3® Polyethylene Insert Study).
Time Frame: Intraoperative
Population: Bone screws used.
Measure: Count of Units; unit: Hips
Units Other Than Participants: Hips
Arm/Group | Tritanium® Primary Acetabular Shell
Number analyzed (Participants) | 234
Number analyzed (Hips) | 241
Hips
  Yes | 178
  No | 63

3. Secondary Outcome: Harris Hip Score
Description: The Harris Hip Score (HHS) assesses pain, function, joint deformity and range of motion. Scores can range from 0 to 100 with 0 being the worst and 100 being the best score. A score of 80-100 is considered good-excellent and a score of less than or equal to 79 is considered fair-poor. 90-100 = excellent 80-89 = good 70-79 = fair 0-69 = poor
Time Frame: 1, 3, and 5 years
Population: A calculable HHS score is a case where all data points are present to calculate the stated score.
Measure: Mean (Standard Deviation); unit: Score on a scale
Units Other Than Participants: Hips
Arm/Group | Tritanium® Primary Acetabular Shell
Number analyzed (Participants) | 234
Number analyzed (Hips) | 241
Score on a scale
  1-Year Harris Hip Score: number analyzed (Participants) | 190
  1-Year Harris Hip Score: number analyzed (Hips) | 192
  1-Year Harris Hip Score | 90.01 (13.6)
  3-Year Harris Hip Score: number analyzed (Participants) | 119
  3-Year Harris Hip Score: number analyzed (Hips) | 122
  3-Year Harris Hip Score | 90.99 (13.64)
  5-Year Harris Hip Score: number analyzed (Participants) | 72
  5-Year Harris Hip Score: number analyzed (Hips) | 74
  5-Year Harris Hip Score | 90.7 (14.37)

4. Secondary Outcome: Short Form- 12 (SF-12) Heath Survey Scores
Description: The SF-12 Health Survey is a 12-item patient completed questionnaire to measure general health and well-being. It includes a physical and mental status component score; each ranging from 0-100. Low values represent a poor health state and high values represent a good health state.
Time Frame: 1, 3, and 5 years
Population: An evaluable case is one where all data points are present to calculate the stated score.
Measure: Mean (Standard Deviation); unit: Score on a scale
Units Other Than Participants: Hips
Arm/Group | Tritanium® Primary Acetabular Shell
Number analyzed (Participants) | 234
Number analyzed (Hips) | 241
Score on a scale
  1-Year Physical Component Score: number analyzed (Participants) | 197
  1-Year Physical Component Score: number analyzed (Hips) | 199
  1-Year Physical Component Score | 46.77 (10.45)
  1-Year Mental Component Score: number analyzed (Participants) | 197
  1-Year Mental Component Score: number analyzed (Hips) | 199
  1-Year Mental Component Score | 55.26 (8.95)
  3-Year Physical Component Score: number analyzed (Participants) | 149
  3-Year Physical Component Score: number analyzed (Hips) | 152
  3-Year Physical Component Score | 46.62 (10.48)
  3-Year Mental Component Score: number analyzed (Participants) | 149
  3-Year Mental Component Score: number analyzed (Hips) | 152
  3-Year Mental Component Score | 55.63 (8.51)
  5-Year Physical Component Score: number analyzed (Participants) | 120
  5-Year Physical Component Score: number analyzed (Hips) | 122
  5-Year Physical Component Score | 46.68 (10.38)
  5-Year Mental Component Score: number analyzed (Participants) | 120
  5-Year Mental Component Score: number analyzed (Hips) | 122
  5-Year Mental Component Score | 55.34 (7.78)

5. Secondary Outcome: Lower Extremity Activity Scale (LEAS) Score
Description: The LEAS is completed by the participant to assess activity level. Activity levels were ordered in terms of intensity from 1 to 18, with 18 indicating the highest activity level.
Time Frame: 1, 3, and 5 years
Population: An evaluable case is one where all data points are present to calculate the stated score.
Measure: Mean (Standard Deviation); unit: Score on a scale
Units Other Than Participants: Hips
Arm/Group | Tritanium® Primary Acetabular Shell
Number analyzed (Participants) | 234
Number analyzed (Hips) | 241
Score on a scale
  1-Year LEAS: number analyzed (Participants) | 200
  1-Year LEAS: number analyzed (Hips) | 202
  1-Year LEAS | 10.74 (3.06)
  3-Year LEAS: number analyzed (Participants) | 149
  3-Year LEAS: number analyzed (Hips) | 152
  3-Year LEAS | 11.61 (3.11)
  5-Year LEAS: number analyzed (Participants) | 120
  5-Year LEAS: number analyzed (Hips) | 122
  5-Year LEAS | 11.11 (3.41)

6. Secondary Outcome: EuroQol Five-Dimensional (EQ-5D)
Description: The EuroQol five-dimensional (EQ-5D) is a subject-completed questionnaire designed to assess subject health state values. The EQ-5D consists of 2 areas: the EQ visual analogue scale (EQ VAS) and EQ-5D descriptive system. The EQ VAS collects health state values using a 20 cm visual analogue scale with the endpoints labeled best imaginable health state at the top and worst imaginable health state at the bottom, having numeric values of 100 to 0 respectively. The EQ-5D Time Trade-off (TTO) descriptive system comprises the following five dimensions: mobility, self-care, usual activities, pain/comfort and anxiety/depression. Each dimension has three levels: no problems, some problems and extreme problems, where an overall score of 1 represents full health.
  The index values on a scale between -1 (low) and 1 (high) are showing the average health status. A low score shows worse health, and a high score shows better health.
Time Frame: 1,2,3,4, and 5 years
Population: A calculable case is one where all data points are present to calculate the stated score.
Measure: Mean (Standard Deviation); unit: Score on a scale
Units Other Than Participants: Hips
Arm/Group | Tritanium® Primary Acetabular Shell
Number analyzed (Participants) | 234
Number analyzed (Hips) | 241
Score on a scale
  1-Year EQ5D Health State Over Time: number analyzed (Participants) | 198
  1-Year EQ5D Health State Over Time: number analyzed (Hips) | 200
  1-Year EQ5D Health State Over Time | 79.87 (17.32)
  1-Year EQ5D TTO Valuation Over Time: number analyzed (Participants) | 200
  1-Year EQ5D TTO Valuation Over Time: number analyzed (Hips) | 202
  1-Year EQ5D TTO Valuation Over Time | .87 (.16)
  2-Year EQ5D Health State Over Time: number analyzed (Participants) | 171
  2-Year EQ5D Health State Over Time: number analyzed (Hips) | 174
  2-Year EQ5D Health State Over Time | 79.87 (17.01)
  2-Year EQ5D TTO Valuation Over Time: number analyzed (Participants) | 171
  2-Year EQ5D TTO Valuation Over Time: number analyzed (Hips) | 174
  2-Year EQ5D TTO Valuation Over Time | .84 (.18)
  3-Year EQ5D Health State Over Time: number analyzed (Participants) | 147
  3-Year EQ5D Health State Over Time: number analyzed (Hips) | 150
  3-Year EQ5D Health State Over Time | 82.75 (13.62)
  3-Year EQ5D TTO Valuation Over Time: number analyzed (Participants) | 147
  3-Year EQ5D TTO Valuation Over Time: number analyzed (Hips) | 150
  3-Year EQ5D TTO Valuation Over Time | .88 (.15)
  4-Year EQ5D Health State Over Time: number analyzed (Participants) | 128
  4-Year EQ5D Health State Over Time: number analyzed (Hips) | 131
  4-Year EQ5D Health State Over Time | 80.8 (15.55)
  4-Year EQ5D TTO Valuation Over Time: number analyzed (Participants) | 128
  4-Year EQ5D TTO Valuation Over Time: number analyzed (Hips) | 131
  4-Year EQ5D TTO Valuation Over Time | .86 (.14)
  5-Year EQ5D Health State Over Time: number analyzed (Participants) | 120
  5-Year EQ5D Health State Over Time: number analyzed (Hips) | 122
  5-Year EQ5D Health State Over Time | 80.95 (16.78)
  5-Year EQ5D TTO Valuation Over Time: number analyzed (Participants) | 120
  5-Year EQ5D TTO Valuation Over Time: number analyzed (Hips) | 122
  5-Year EQ5D TTO Valuation Over Time | .86 (.15)

7. Secondary Outcome: Follow-Up Questionnaire
Description: The Follow-up Questionnaire is a short patient questionnaire intended to provide information on patient satisfaction, pain, and whether or not there have been any revisions or removals since the last follow-up visit. It consists of three questions:
  * Patient satisfaction with the hip replacement
  * Presence of any pain in the study hip
  * Any surgeries performed on the study hip
Time Frame: 6, 7, 8, 9, and 10 years
Population: Not all participants completed the Follow-Up Questionnaire at the respective timepoints.
Measure: Count of Units; unit: Hips
Units Other Than Participants: Hips
Arm/Group | Tritanium® Primary Acetabular Shell
Number analyzed (Participants) | 234
Number analyzed (Hips) | 241
Hips
  6-Year_ Follow-up Questionnaire _Q1: Pain in Study Hip? - YES: number analyzed (Participants) | 97
  6-Year_ Follow-up Questionnaire _Q1: Pain in Study Hip? - YES: number analyzed (Hips) | 99
  6-Year_ Follow-up Questionnaire _Q1: Pain in Study Hip? - YES | 25
  6-Year_ Follow-up Questionnaire _Q1: Pain in Study Hip? - NO: number analyzed (Participants) | 97
  6-Year_ Follow-up Questionnaire _Q1: Pain in Study Hip? - NO: number analyzed (Hips) | 99
  6-Year_ Follow-up Questionnaire _Q1: Pain in Study Hip? - NO | 74
  6-Year_Follow-up Questionnaire_Q2: Satisfied with Results of Hip Replacement? - YES: number analyzed (Participants) | 97
  6-Year_Follow-up Questionnaire_Q2: Satisfied with Results of Hip Replacement? - YES: number analyzed (Hips) | 99
  6-Year_Follow-up Questionnaire_Q2: Satisfied with Results of Hip Replacement? - YES | 96
  6-Year_Follow-up Questionnaire_Q2: Satisfied with Results of Hip Replacement? - NO: number analyzed (Participants) | 97
  6-Year_Follow-up Questionnaire_Q2: Satisfied with Results of Hip Replacement? - NO: number analyzed (Hips) | 99
  6-Year_Follow-up Questionnaire_Q2: Satisfied with Results of Hip Replacement? - NO | 3
  6-Year_Follow-up Questionnaire_Q3: Surgery on Study Hip Since Last Study visit? - YES: number analyzed (Participants) | 97
  6-Year_Follow-up Questionnaire_Q3: Surgery on Study Hip Since Last Study visit? - YES: number analyzed (Hips) | 99
  6-Year_Follow-up Questionnaire_Q3: Surgery on Study Hip Since Last Study visit? - YES | 1
  6-Year_Follow-up Questionnaire_Q3: Surgery on Study Hip Since Last Study visit? - NO: number analyzed (Participants) | 97
  6-Year_Follow-up Questionnaire_Q3: Surgery on Study Hip Since Last Study visit? - NO: number analyzed (Hips) | 99
  6-Year_Follow-up Questionnaire_Q3: Surgery on Study Hip Since Last Study visit? - NO | 98
  7-Year_ Follow-up Questionnaire _Q1: Pain in Study Hip? - YES: number analyzed (Participants) | 87
  7-Year_ Follow-up Questionnaire _Q1: Pain in Study Hip? - YES: number analyzed (Hips) | 89
  7-Year_ Follow-up Questionnaire _Q1: Pain in Study Hip? - YES | 25
  7-Year_ Follow-up Questionnaire _Q1: Pain in Study Hip? - NO: number analyzed (Participants) | 87
  7-Year_ Follow-up Questionnaire _Q1: Pain in Study Hip? - NO: number analyzed (Hips) | 89
  7-Year_ Follow-up Questionnaire _Q1: Pain in Study Hip? - NO | 64
  7-Year_Follow-up Questionnaire_Q2: Satisfied with Results of Hip Replacement? - YES: number analyzed (Participants) | 87
  7-Year_Follow-up Questionnaire_Q2: Satisfied with Results of Hip Replacement? - YES: number analyzed (Hips) | 89
  7-Year_Follow-up Questionnaire_Q2: Satisfied with Results of Hip Replacement? - YES | 86
  7-Year_Follow-up Questionnaire_Q2: Satisfied with Results of Hip Replacement? - NO: number analyzed (Participants) | 87
  7-Year_Follow-up Questionnaire_Q2: Satisfied with Results of Hip Replacement? - NO: number analyzed (Hips) | 89
  7-Year_Follow-up Questionnaire_Q2: Satisfied with Results of Hip Replacement? - NO | 3
  7-Year_Follow-up Questionnaire_Q3: Surgery on Study Hip Since Last Study visit? - YES: number analyzed (Participants) | 87
  7-Year_Follow-up Questionnaire_Q3: Surgery on Study Hip Since Last Study visit? - YES: number analyzed (Hips) | 89
  7-Year_Follow-up Questionnaire_Q3: Surgery on Study Hip Since Last Study visit? - YES | 0
  7-Year_Follow-up Questionnaire_Q3: Surgery on Study Hip Since Last Study visit? - NO: number analyzed (Participants) | 87
  7-Year_Follow-up Questionnaire_Q3: Surgery on Study Hip Since Last Study visit? - NO: number analyzed (Hips) | 89
  7-Year_Follow-up Questionnaire_Q3: Surgery on Study Hip Since Last Study visit? - NO | 89
  8-Year_ Follow-up Questionnaire _Q1: Pain in Study Hip? - YES: number analyzed (Participants) | 63
  8-Year_ Follow-up Questionnaire _Q1: Pain in Study Hip? - YES: number analyzed (Hips) | 64
  8-Year_ Follow-up Questionnaire _Q1: Pain in Study Hip? - YES | 14
  8-Year_ Follow-up Questionnaire _Q1: Pain in Study Hip? - NO: number analyzed (Participants) | 63
  8-Year_ Follow-up Questionnaire _Q1: Pain in Study Hip? - NO: number analyzed (Hips) | 64
  8-Year_ Follow-up Questionnaire _Q1: Pain in Study Hip? - NO | 50
  8-Year_Follow-up Questionnaire_Q2: Satisfied with Results of Hip Replacement? - YES: number analyzed (Participants) | 63
  8-Year_Follow-up Questionnaire_Q2: Satisfied with Results of Hip Replacement? - YES: number analyzed (Hips) | 64
  8-Year_Follow-up Questionnaire_Q2: Satisfied with Results of Hip Replacement? - YES | 61
  8-Year_Follow-up Questionnaire_Q2: Satisfied with Results of Hip Replacement? - NO: number analyzed (Participants) | 63
  8-Year_Follow-up Questionnaire_Q2: Satisfied with Results of Hip Replacement? - NO: number analyzed (Hips) | 64
  8-Year_Follow-up Questionnaire_Q2: Satisfied with Results of Hip Replacement? - NO | 3
  8-Year_Follow-up Questionnaire_Q3: Surgery on Study Hip Since Last Study visit? - YES: number analyzed (Participants) | 63
  8-Year_Follow-up Questionnaire_Q3: Surgery on Study Hip Since Last Study visit? - YES: number analyzed (Hips) | 64
  8-Year_Follow-up Questionnaire_Q3: Surgery on Study Hip Since Last Study visit? - YES | 0
  8-Year_Follow-up Questionnaire_Q3: Surgery on Study Hip Since Last Study visit? - NO: number analyzed (Participants) | 63
  8-Year_Follow-up Questionnaire_Q3: Surgery on Study Hip Since Last Study visit? - NO: number analyzed (Hips) | 64
  8-Year_Follow-up Questionnaire_Q3: Surgery on Study Hip Since Last Study visit? - NO | 64
  9-Year_ Follow-up Questionnaire _Q1: Pain in Study Hip? - YES: number analyzed (Participants) | 39
  9-Year_ Follow-up Questionnaire _Q1: Pain in Study Hip? - YES: number analyzed (Hips) | 39
  9-Year_ Follow-up Questionnaire _Q1: Pain in Study Hip? - YES | 8
  9-Year_ Follow-up Questionnaire _Q1: Pain in Study Hip? - NO: number analyzed (Participants) | 39
  9-Year_ Follow-up Questionnaire _Q1: Pain in Study Hip? - NO: number analyzed (Hips) | 39
  9-Year_ Follow-up Questionnaire _Q1: Pain in Study Hip? - NO | 31
  9-Year_Follow-up Questionnaire_Q2: Satisfied with Results of Hip Replacement? - YES: number analyzed (Participants) | 39
  9-Year_Follow-up Questionnaire_Q2: Satisfied with Results of Hip Replacement? - YES: number analyzed (Hips) | 39
  9-Year_Follow-up Questionnaire_Q2: Satisfied with Results of Hip Replacement? - YES | 38
  9-Year_Follow-up Questionnaire_Q2: Satisfied with Results of Hip Replacement? - NO: number analyzed (Participants) | 39
  9-Year_Follow-up Questionnaire_Q2: Satisfied with Results of Hip Replacement? - NO: number analyzed (Hips) | 39
  9-Year_Follow-up Questionnaire_Q2: Satisfied with Results of Hip Replacement? - NO | 1
  9-Year_Follow-up Questionnaire_Q3: Surgery on Study Hip Since Last Study visit? - YES: number analyzed (Participants) | 39
  9-Year_Follow-up Questionnaire_Q3: Surgery on Study Hip Since Last Study visit? - YES: number analyzed (Hips) | 39
  9-Year_Follow-up Questionnaire_Q3: Surgery on Study Hip Since Last Study visit? - YES | 0
  9-Year_Follow-up Questionnaire_Q3: Surgery on Study Hip Since Last Study visit? - NO: number analyzed (Participants) | 39
  9-Year_Follow-up Questionnaire_Q3: Surgery on Study Hip Since Last Study visit? - NO: number analyzed (Hips) | 39
  9-Year_Follow-up Questionnaire_Q3: Surgery on Study Hip Since Last Study visit? - NO | 39
  10-Year_ Follow-up Questionnaire _Q1: Pain in Study Hip? - YES: number analyzed (Participants) | 41
  10-Year_ Follow-up Questionnaire _Q1: Pain in Study Hip? - YES: number analyzed (Hips) | 43
  10-Year_ Follow-up Questionnaire _Q1: Pain in Study Hip? - YES | 6
  10-Year_ Follow-up Questionnaire _Q1: Pain in Study Hip? - NO: number analyzed (Participants) | 41
  10-Year_ Follow-up Questionnaire _Q1: Pain in Study Hip? - NO: number analyzed (Hips) | 43
  10-Year_ Follow-up Questionnaire _Q1: Pain in Study Hip? - NO | 37
  10-Year_Follow-up Questionnaire_Q2: Satisfied with Results of Hip Replacement? - YES: number analyzed (Participants) | 41
  10-Year_Follow-up Questionnaire_Q2: Satisfied with Results of Hip Replacement? - YES: number analyzed (Hips) | 43
  10-Year_Follow-up Questionnaire_Q2: Satisfied with Results of Hip Replacement? - YES | 41
  10-Year_Follow-up Questionnaire_Q2: Satisfied with Results of Hip Replacement? - NO: number analyzed (Participants) | 41
  10-Year_Follow-up Questionnaire_Q2: Satisfied with Results of Hip Replacement? - NO: number analyzed (Hips) | 43
  10-Year_Follow-up Questionnaire_Q2: Satisfied with Results of Hip Replacement? - NO | 2
  10-Year_Follow-up Questionnaire_Q3: Surgery on Study Hip Since Last Study visit? - YES: number analyzed (Participants) | 41
  10-Year_Follow-up Questionnaire_Q3: Surgery on Study Hip Since Last Study visit? - YES: number analyzed (Hips) | 43
  10-Year_Follow-up Questionnaire_Q3: Surgery on Study Hip Since Last Study visit? - YES | 0
  10-Year_Follow-up Questionnaire_Q3: Surgery on Study Hip Since Last Study visit? - NO: number analyzed (Participants) | 41
  10-Year_Follow-up Questionnaire_Q3: Surgery on Study Hip Since Last Study visit? - NO: number analyzed (Hips) | 43
  10-Year_Follow-up Questionnaire_Q3: Surgery on Study Hip Since Last Study visit? - NO | 43

8. Secondary Outcome: Acetabular Shell Radiographic Stability
Description: Numerous parameters will be reviewed by zone, including radiolucency and migration. All data will be evaluated in order to classify each case as stable or unstable.
Time Frame: 6 weeks, 1, 3, 5 years
Population: Frequency of the acetabular shell stability.
Measure: Count of Units; unit: Hips
Units Other Than Participants: Hips
Arm/Group | Tritanium® Primary Acetabular Shell
Number analyzed (Participants) | 234
Number analyzed (Hips) | 241
Hips
  6- Weeks Postoperative: Stable: number analyzed (Participants) | 222
  6- Weeks Postoperative: Stable: number analyzed (Hips) | 227
  6- Weeks Postoperative: Stable | 227
  6- Weeks Postoperative: Fibrous Stable: number analyzed (Participants) | 222
  6- Weeks Postoperative: Fibrous Stable: number analyzed (Hips) | 227
  6- Weeks Postoperative: Fibrous Stable | 0
  6- Weeks Postoperative: Unstable: number analyzed (Participants) | 222
  6- Weeks Postoperative: Unstable: number analyzed (Hips) | 227
  6- Weeks Postoperative: Unstable | 0
  1-Year Postoperative: Stable: number analyzed (Participants) | 191
  1-Year Postoperative: Stable: number analyzed (Hips) | 194
  1-Year Postoperative: Stable | 192
  1-Year Postoperative: Fibrous Stable: number analyzed (Participants) | 191
  1-Year Postoperative: Fibrous Stable: number analyzed (Hips) | 194
  1-Year Postoperative: Fibrous Stable | 2
  1-Year Postoperative: Unstable: number analyzed (Participants) | 191
  1-Year Postoperative: Unstable: number analyzed (Hips) | 194
  1-Year Postoperative: Unstable | 0
  3-Years Postoperative: Stable: number analyzed (Participants) | 131
  3-Years Postoperative: Stable: number analyzed (Hips) | 134
  3-Years Postoperative: Stable | 130
  3-Years Postoperative: Fibrous Stable: number analyzed (Participants) | 131
  3-Years Postoperative: Fibrous Stable: number analyzed (Hips) | 134
  3-Years Postoperative: Fibrous Stable | 4
  3-Years Postoperative: Unstable: number analyzed (Participants) | 131
  3-Years Postoperative: Unstable: number analyzed (Hips) | 134
  3-Years Postoperative: Unstable | 0
  5-Years Postoperative: Stable: number analyzed (Participants) | 89
  5-Years Postoperative: Stable: number analyzed (Hips) | 91
  5-Years Postoperative: Stable | 85
  5-Years Postoperative: Fibrous Stable: number analyzed (Participants) | 89
  5-Years Postoperative: Fibrous Stable: number analyzed (Hips) | 91
  5-Years Postoperative: Fibrous Stable | 3
  5-Years Postoperative: Unstable: number analyzed (Participants) | 89
  5-Years Postoperative: Unstable: number analyzed (Hips) | 91
  5-Years Postoperative: Unstable | 3

ADVERSE EVENTS:
Time Frame: Participants were assessed up to 10 years.
Description: Censored cases were not included as at risk. Date of occurrence, date diagnosed, type of complication and treatment were collected. Industry standard adverse events (AE) and serious adverse events (SAE) terms were used in this study.
Groups:
- Operative Site Adverse Event(s): Operative site adverse events are reported by study hip because in the case of bilateral participants (participants who have the study device implanted in both hips), an event can occur in one hip, both hips or the same hip, but at different times and are counted as separate events for this reason.
- Non-operative Site Adverse Event(s): Non-operative site adverse events that were reported by participant.
Arm/Group | Operative Site Adverse Event(s) | Non-operative Site Adverse Event(s)
All-Cause Mortality (participants affected / at risk) | 0/241 | 13/234
Serious Adverse Events (participants affected / at risk) | 16/241 | 56/234
Other Adverse Events (participants affected / at risk) | 61/241 | 0/234
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Operative Site Adverse Event(s) (N=241) | Non-operative Site Adverse Event(s) (N=234)
Operative Site (Infections and infestations) | 6 (6) | 0 (0) — Deep Joint Infection; Superficial Wound Infection
Operative Site (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) — Wound Hematoma
Operative Site (Musculoskeletal and connective tissue disorders) | 7 (9) | 0 (0) — Acetabular Component Loosening; Femoral Component Loosening, Hip Pain, Femoral Crack Fracture, Trauma, Tibial Plateau Fracture
Non-Operative (Blood and lymphatic system disorders) | 0 (0) | 2 (3) — Anemia; Hemolytic Anemia
Non-Operative (Cardiac disorders) | 0 (0) | 17 (19) — AV Block; A-FIB; NSTEMI; Abdominal Aortic Aneurysm; Angina / Acute Coronary Syndrome; Unstable Angina Pectoris; HTN; Exacerbation of CHF; CHF; Pacemaker Implant; HTN Crisis; Symptomatic Bradycardia with Hypotension; Vertigo; MI; Microcytic Anemia
Non-Operative (Eye disorders) | 0 (0) | 1 (1) — R-Eye Retinal Detachment
Non-operative (Gastrointestinal disorders) | 0 (0) | 5 (7) — Ischemic Colitis; Cholecystitis; Mild Postoperative Ileus; Partial SBO; Partial Bowel Obstruction; Small Bowel Obstruction; Acute Colitis and Leukocytosis
Non-Operative (General disorders) | 0 (0) | 4 (4) — Death (cause unspecified); vertigo
Non-Operative (Hepatobiliary disorders) | 0 (0) | 1 (1) — Acute Cholecystitis
Non-Operative (Infections and infestations) | 0 (0) | 2 (2) — Pneumonia; Infection; Urinary Tract Infection; Pneumonia, Acute Exacerbation of COPD
Non-Operative (Musculoskeletal and connective tissue disorders) | 0 (0) | 12 (13) — Herniated Disk; Tibial & Fibula Fractures, Sprained Muscle; Trauma; Lumbar Pain; Hip OA; Spinal Stenosis; Scoliosis; Herniated Nucleus Pulposus; Spondylosis; Knee OA; Lumbar/Lateral Recess Stenosis; MVC, Polytrauma; Rib Fractures; Subscap Hematoma
Non-Operative (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 14 (17) — Breast; Colon; Osteosarcoma and Metastatic Osteosarcoma; Sarcoma; Leiomyosarcoma; Squamous Cell, Prostate; GI malignancy; Pituitary Adenoma
Non-Operative (Nervous system disorders) | 0 (0) | 7 (10) — Neuropathy; Lower Extremity Weakness; Altered Mental Status; Headaches; Aneurysm; Disorientation and Memory Loss; Idiopathic Tremor; Encephalopathy, Cognitive Decline
Non-operative (Psychiatric disorders) | 0 (0) | 1 (1) — Alcoholism
Non-Operative (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (8) — COPD; Exacerbation of COPD; Anaphylactic Shock (Insect Sting); Choked
Non-Operative (Surgical and medical procedures) | 0 (0) | 1 (1) — Evacuation of hematoma and removal of extruded herniated nucleus pulposus and endplate cartilage.
Non-Operative (Vascular disorders) | 0 (0) | 8 (8) — DVT; Pulmonary Embolism; Cerebrovascular Accident, Stroke, Aneurysm
Non-Operative (Renal and urinary disorders) | 0 (0) | 1 (1) — Urinary tract infection
Operative (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) — Femoral osteosarcoma
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Operative Site Adverse Event(s) (N=241) | Non-operative Site Adverse Event(s) (N=234)
Operative Site (Musculoskeletal and connective tissue disorders) | 61 (90) | 0 — Tendonitis; Bursitis; Hip Pain; Soft Tissue Trauma; Groin Pain: Neuritis; Acetabular Component Loosening; Femoral Crack fracture

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There is an agreement between Principal Investigators and the Sponsor (or its agents) that requires Investigators to allow Sponsor at least 30 days to review material intended for publications in order to redact any Confidential Information or Inventions therefrom.

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-08-24): https://cdn.clinicaltrials.gov/large-docs/51/NCT01063751/Prot_SAP_ICF_000.pdf